CLINICAL TRIAL: NCT05418153
Title: Evaluating the New Synergy IOL - First 7 Months Data From Two US Centers
Brief Title: Synergy Lens Outcomes Evaluation
Status: Completed | Type: Observational
Sponsor: Center For Sight (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Other Study IDs: CFS 21-001
Record Dates: First submitted 2022-06-08; First posted 2022-06-14 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2022-06

CONDITIONS: Presbyopia; Pseudophakia
MeSH Terms: conditions — Presbyopia; Pseudophakia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Synergy IOL: Patients implanted with the Synergy IOL in both eyes.
  Interventions: Device: Tecnis Synergy IOL

INTERVENTIONS:
Device: Tecnis Synergy IOL — Intraocular lens replaces the natural lens removed during cataract surgery in both eyes.

SUMMARY:
This is a single visit study to evaluate the visual outcomes and patient satisfaction of patients who were bilaterally implanted with the Tecnis Synergy IOL between June 1 and December 31, 2021 in 2 centers in USA

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Gender: Males and Females.
3. Uneventful bilateral lens extraction
4. Bilateral implantation of Synergy IOLs (toric and non-toric) by 5 anterior segment surgeons at Center For Sight (DWS, WJL, JWK, WLS, and JOD) and 1 surgeon at Carolina Eyecare Physicians (KDS) through the months of June to December 2021.
5. Willing and able to provide written informed consent for participation in the study.
6. Willing and able to comply with scheduled visit and study examination procedures.
7. At least 3 months postoperative from second eye IOL implantation.
8. Postoperative best corrected visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

1. Established ocular pathology, including: glaucoma (except glaucoma suspects), uveitis, and clinically-significant retinal pathology affecting the macula (with visual acuity worse than 20/32) and/or any other ocular findings that may, in the opinion of the investigator, affect vision.
2. Uncontrolled diabetes.
3. Use of any systemic or topical drug known to interfere with visual performance.
4. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
5. Clinically significant corneal dystrophy.
6. Irregular astigmatism.
7. History of chronic intraocular inflammation.
8. Previous intraocular surgery.
9. Previous keratoplasty
10. Previous refractive surgery.
11. Severe dry eye
12. Pupil abnormalities
13. Any clinically significant, serious or severe medical or psychiatric condition that may interfere with the interpretation of study results.
14. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.
15. Best-corrected distance visual acuity worse than 20/32 in each eye.
16. Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
17. Abnormal iris
18. Patients who had a complication during cataract surgery, which could include ruptured zonules, torn capsule, or vitrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent routine, uneventful cataract surgery with implantation of the Synergy lens in both eyes between 01June2021 and 31Dec2021 at Center For Sight (Sarasota, FL) and Carolina Eyecare Physicians (Charleston, SC)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center For Sight, Venice, Florida
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synergy IOL
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Synergy IOL
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 45
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance Corrected Near Visual Acuity at 40 cm Under Photopic Conditions
Description: Visual acuity measured at 40 cm
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Synergy IOL
Number analyzed (Participants) | 52
logMAR | 0.01 (0.07)

2. Primary Outcome: Binocular Distance Corrected Near Visual Acuity at 40 cm Under Mesopic Conditions
Description: Visual acuity measured at 40 cm under dim light
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Synergy IOL
Number analyzed (Participants) | 35
logMAR | 0.21 (0.12)

ADVERSE EVENTS:
Time Frame: Day of study visit
Arm/Group | Synergy IOL
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT05418153/Prot_SAP_000.pdf